CLINICAL TRIAL: NCT03891446
Title: An Extension Trial to Evaluate the Long-term Safety and Efficacy of Bimatoprost SR in Patients With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Long-term Safety and Efficacy Extension Trial of Bimatoprost SR
Acronym: MAIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1698-302-007; 2018-003597-26 (EudraCT Number); 2023-504601-36-00 (Other: EU CT)
Expanded Access: NCT05338606 (No longer available)
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension; Bimatoprost; DURYSTA
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lead-in study 192024-091 or -092 or -095 (Experimental): Study eye (Eye that received Bimatoprost SR in the lead-in study): No treatment is administered.
  Fellow eye (Eye that did not receive Bimatoprost SR in the lead-in study): Fellow eye will receive only standard of care, based on the investigator's judgment.
  Interventions: Other: Standard of Care
- Lead-in study 192024-093 Stage 1 (Experimental): Participants who received 1, 2 or 3 administrations and participants in Stage 2 who received 1 Bimatoprost SR administration due to safety concern or received 2 administrations.
  Study eye (Eye that received Bimatoprost SR in the lead-in study): No treatment is administered.
  Fellow eye (Eye that did not receive Bimatoprost SR in the lead-in study): Fellow eye will receive only standard of care, based on the investigator's judgment.
  Interventions: Other: Standard of Care
- Lead-in study 192024-093 Stage 2 (Experimental): Participants who received 1 Bimatoprost administration due to sustained efficacy:
  Study eye (Eye that received Bimatoprost SR in the lead-in study): 1 additional administration of Bimatoprost SR may be administered through completion of the Month 12 visit, at least 4 months apart from the lead-in study administration. Fellow eye (Eye that did not receive Bimatoprost SR in the lead-in study): Fellow eye will receive only standard of care, based on the investigator's judgment.
  Interventions: Drug: Bimatoprost SR; Other: Standard of Care
- Lead-in study ARGOS (Experimental): Study eye (Eye that received Bimatoprost SR first in the lead-in study): 1 additional administration of Bimatoprost SR may be administered through completion of the Month 12 visit, at least 4 months apart from the lead-in study administration.
  Treated Fellow eye (Eye that received Bimatoprost SR second in the lead-in study): 1 additional administration of Bimatoprost SR may be administered through completion of the Month 12 visit, at least 4 months apart from the lead-in study administration.
  Untreated Fellow eye (Eye that did not receive Bimatoprost SR in the lead-in study): Untreated fellow eye will receive only standard of care, based on the investigator's judgment.
  Interventions: Drug: Bimatoprost SR; Other: Standard of Care

INTERVENTIONS:
Drug: Bimatoprost SR — Intraocular implant
  Other Names: DURYSTA
  Arms: Lead-in study 192024-093 Stage 2; Lead-in study ARGOS
Other: Standard of Care — Standard of care treatment based on investigator's judgement.

SUMMARY:
This study will evaluate the long-term safety and efficacy of Bimatoprost Sustained Release (SR) in patients with open-angle glaucoma or ocular hypertension who completed 1 of the 4 Phase 3 Bimatoprost SR studies (192024-091, -092, -093, or -095) and received Bimatoprost SR or who received commercial DURYSTA (Bimatoprost SR) in the open-label Phase 4 ARGOS study (MED-MA-EYE-0648) and completed (or exited early from) the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed 1 of the 4 Bimatoprost SR Phase 3 studies (192024-091, -092, -093, or -095) and received Bimatoprost SR.
* Participants who completed (or exited early from) the open-label Phase 4 ARGOS study with no ongoing safety concerns, and received DURYSTA.

Exclusion Criteria:

* Female participants who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using a reliable means of contraception during the study.
* Concurrent or anticipated enrollment in another investigational drug or device study during the present study.
* Any condition which would preclude the participant's ability to comply with study requirements, including completion of the study.
* Participants who were randomized to receive timolol eye drops in the study eye (control group) during the Phase 3 Bimatoprost Studies 192024-091 and -092.
* For patients from the ARGOS lead-in study: history of prior incisional glaucoma surgeries and/or minimally invasive glaucoma surgical procedures in the study eye or treated fellow eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Duration of effect of Bimatoprost SR | Approximately 24 months
  Retreatment or rescue administered for IOP lowering, determined by the investigator.
Number of patients experiencing a treatment emergent adverse event | Approximately 24 months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (124):
- United States (66):
  - Trinity Research Group /ID# 240190, Dothan, Alabama
  - Arizona Eye Center - West Ray Road /ID# 240239, Chandler, Arizona
  - Arizona Glaucoma Specialists /ID# 240212, Phoenix, Arizona
  - M&M Eye Institute /ID# 240236, Prescott, Arizona
  - Horizon Eye Specialists & Lasik Centers /ID# 240255, Sun City, Arizona
  - Angeles Eye Institute /ID# 250397, Culver City, California
  - Duplicate_Lakeside Vision Center /ID# 240204, Irvine, California
  - Hamilton Glaucoma Center Shiley Eye Center UCSD /ID# 240196, La Jolla, California
  - The Eye Research Foundation /ID# 240186, Newport Beach, California
  - North Bay Eye Associates Inc. /ID# 248912, Petaluma, California
  - Duplicate_Martel Eye Medical Group /ID# 240291, Rancho Cordova, California
  - The Clinical Trials Network (CTNx) /ID# 240284, Redding, California
  - Sacramento Eye Consultants /ID# 240263, Sacramento, California
  - Pacific Eye Associates /ID# 240234, San Francisco, California
  - Wolstan & Goldberg Eye Associates /ID# 240221, Torrance, California
  - Colorado Eye Institute /ID# 248910, Colorado Springs, Colorado
  - Specialty Retina Center /ID# 240254, Coral Springs, Florida
  - Nature Coast Clinical Research - Crystal River /ID# 240334, Crystal River, Florida
  - Bruce Segal, MD /ID# 240292, Delray Beach, Florida
  - Eye Associates of Fort Meyers /ID# 240218, Fort Myers, Florida
  - Levenson Eye Associates Inc. /ID# 240209, Jacksonville, Florida
  - MedEye Associates /ID# 240333, Miami, Florida
  - Logan Ophthalmic Research Inc. /ID# 240280, Tamarac, Florida
  - International Research Center /ID# 240346, Tampa, Florida
  - University of South Florida- Neuroscience Institute /ID# 250980, Tampa, Florida
  - Duplicate_Emory University /ID# 240328, Atlanta, Georgia
  - Coastal Research Associates /ID# 240192, Roswell, Georgia
  - Chicago Eye Specialists /ID# 240270, Bedford Park, Illinois
  - University of Illinois at Chicago /ID# 250981, Chicago, Illinois
  - Kovach Eye Institute /ID# 250442, Elmhurst, Illinois
  - IN Univ School of Medicine /ID# 240294, Indianapolis, Indiana
  - The Eye Care Institute /ID# 240289, Louisville, Kentucky
  - Duplicate_Tulane University /ID# 240327, New Orleans, Louisiana
  - Clinical Eye Research of Boston LLC /ID# 240203, Winchester, Massachusetts
  - Fraser Eye Center /ID# 240245, Fraser, Michigan
  - Midwest Vision Research Foundation at Pepose Vision Institute /ID# 250402, Chesterfield, Missouri
  - Tekwani Vision Center /ID# 240220, St Louis, Missouri
  - Eye Associates of North Jersey /ID# 250445, Dover, New Jersey
  - Glaucoma Care Center /ID# 250978, Livingston, New Jersey
  - Rutgers New Jersey Medical School Campus, Doctors Office Center /ID# 240181, Newark, New Jersey
  - Eye Associates of New Mexico /ID# 240216, Albuquerque, New Mexico
  - Ophthalmic Consultants Long Island /ID# 240211, Oceanside, New York
  - Rochester Ophthalmological Group PC /ID# 240290, Rochester, New York
  - Glaucoma associates/consultants of the capital region /ID# 240195, Slingerlands, New York
  - Montefiore Hospital /ID# 240324, The Bronx, New York
  - Asheville Eye Associates /ID# 240202, Asheville, North Carolina
  - Charlotte Eye,Ear,Nose Throat /ID# 240339, Belmont, North Carolina
  - Albemarle Clinical Trials LLC /ID# 240219, Elizabeth City, North Carolina
  - Private Practice - Dr. James D. Branch /ID# 240188, Winston-Salem, North Carolina
  - Bergstrom Eye Research LLC /ID# 240257, Fargo, North Dakota
  - Oklahoma Eye Surgeons /ID# 250430, Oklahoma City, Oklahoma
  - Legacy Devers Eye Institute /ID# 240210, Portland, Oregon
  - Scott and Christie and Associates /ID# 240189, Cranberry Township, Pennsylvania
  - Eye Specialty Group /ID# 240241, Memphis, Tennessee
  - Vanderbilt Eye Institute /ID# 252659, Nashville, Tennessee
  - Advancing Vision Research /ID# 240288, Smyrna, Tennessee
  - Keystone Research LTD /ID# 240185, Austin, Texas
  - Houston Eye Associates /ID# 240340, Houston, Texas
  - DCT Shah Eye Research Institut /ID# 240306, Mission, Texas
  - Plano Office /ID# 240243, Plano, Texas
  - San Antonio Eye Center /ID# 240238, San Antonio, Texas
  - Eye associates /ID# 240265, San Antonio, Texas
  - Medical Center Ophthalmology Associates /ID# 240208, San Antonio, Texas
  - Emerson Clinical Research Institute. LLC /ID# 240274, Falls Church, Virginia
  - Piedmont Eye Center /ID# 240187, Lynchburg, Virginia
  - Vistar Eye Center /ID# 240198, Roanoke, Virginia
- Argentina (5):
  - Consultorio Oftalmologico Dr. Fabian Lerner /ID# 240247, CABA, Buenos Aires
  - Clinica Privada de Ojos /ID# 240272, Mar del Plata, Buenos Aires
  - Hospital Universitario Austral /ID# 240331, Pilar, Buenos Aires
  - Oftalmología Global /ID# 240244, Rosario, Santa Fe Province
  - Oftar Mendoza /ID# 240308, Mendoza
- Universitair Ziekenhuis Leuven /ID# 240312, Leuven, Vlaams-Brabant, Belgium
- Brazil (4):
  - Hospital de Olhos de Mato Grosso Do Sul /ID# 240276, Campo Grande, Mato Grosso do Sul
  - Clinica De Oftalmologia Nova Campinas /ID# 240271, Campinas, São Paulo
  - Hospital Oftalmologico Medicina dos Olhos /ID# 240277, Osasco, São Paulo
  - Hospital Sao Paulo /ID# 240278, São Paulo
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre - Victoria General /ID# 240336, Halifax, Nova Scotia
  - Ophthalmic Consultant Centres /ID# 240205, Mississauga, Ontario
- Colombia (3):
  - Clinica de Oftalmologia Sandiego /ID# 240233, Medellín, Antioquia
  - Fundacion Oftalmologica Nacional /ID# 240226, Bogotá, Bogota D.C.
  - Fundacion Oftalmologica de Santander - FOSCAL /ID# 240634, Bucaramanga, Santander Department
- Ocni klinika Pardubice /ID# 240347, Pardubice, Czechia
- Rigshospitalet Glostrup /ID# 240330, Glostrup Municipality, Capital Region, Denmark
- Egypt (2):
  - Bostan Diagnostic Eye Center /ID# 240268, Cairo
  - Duplicate_Ain Shams University Hospital /ID# 240338, Cairo
- France (2):
  - CHU Bordeaux - Hopital Pellegrin /ID# 240316, Bordeaux, Nouvelle-Aquitaine
  - Centre Ophtalmologique Pôle Vision /ID# 240256, Écully, Rhone
- Germany (2):
  - Internationale Innovative Ophthalmochirurgie /ID# 240232, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Magdeburg /ID# 240314, Magdeburg
- The Chinese University of Hong Kong /ID# 240283, Hong Kong, Hong Kong
- Israel (5):
  - Galilee Medical Center /ID# 251967, Nahariya, Northern District
  - Tel Aviv Sourasky Medical Center /ID# 240311, Tel Aviv, Tel Aviv
  - Rambam Health Care Campus /ID# 240332, Haifa
  - Bnai Zion Medical Center /ID# 240297, Haifa
  - The Lady Davis Carmel Medical Center /ID# 240293, Haifa
- Italy (4):
  - AOU Policlinico G. Rodolico - San Marco /ID# 240305, Catania
  - ASL 2 Abruzzo Lanciano-Vasto-Chieti /ID# 240217, Chieti
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia /ID# 240310, Perugia
  - Azienda Ospedaliero Universitaria Pisana /ID# 240301, Pisa
- Capital Eye Specialists /ID# 240259, Wellington, New Zealand
- Centro Oftalmologico Macula Diagnostico and Tratamiento /ID# 240269, Lima, Peru
- Philippines (3):
  - Asian Eye Institute /ID# 240213, Makati City
  - Asian Eye Institute /ID# 240214, Makati City
  - Peregrine Eye and Laser Institute /ID# 240260, Makati City
- Poland (4):
  - Oftalmika sp. z o.o. /ID# 240201, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Klinika Diagnostyki i Mikrochirurgii Jaskry /ID# 240258, Lublin, Lublin Voivodeship
  - Duplicate_Optimum Profesorskie Centrum Okulistyki Sp. z o.o. /ID# 240307, Gdansk, Pomeranian Voivodeship
  - Centrum Diagnostyki i Mikrochirurgii Oka - LENS sp. z o.o /ID# 240248, Olsztyn, Warmian-Masurian Voivodeship
- Russia (2):
  - S. Fyodorov Eye Microsurgery Federal State Institution /ID# 240251, Novosibirsk, Novosibirsk Oblast
  - Clinical ophthalmology hospital n.a. V.P. Vihodtsev. /ID# 240253, Omsk, Omsk Oblast
- Singapore National Eye Centre /ID# 240224, Singapore, Singapore
- Pretoria Eye Institute - Private Practice /ID# 240223, Pretoria, Gauteng, South Africa
- South Korea (3):
  - Asan Medical Center /ID# 240286, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 240335, Seoul, Seoul Teugbyeolsi
  - Duplicate_Seoul National University Hospital /ID# 240262, Seoul
- Spain (3):
  - Hospital Universitario Reina Sofia /ID# 240322, Córdoba, Cordoba
  - Hospital Clinico San Carlos /ID# 240303, Madrid
  - Hospital Universitario Virgen Macarena /ID# 240325, Seville
- Thailand (2):
  - Maharaj Nakorn Chiang Mai Hospital /ID# 240194, Chiang Mai
  - Thammasat University Hospital /ID# 240231, Pathum Thani
- Turkey (Türkiye) (2):
  - Eskisehir Osmangazi University Medical School /ID# 240225, Eskişehir
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi /ID# 240296, Istanbul
- United Kingdom (2):
  - Addenbrookes Hospital /ID# 240351, Cambridge, Cambridgeshire
  - Duplicate_NHS Lothian /ID# 240318, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=1698-302-007